CLINICAL TRIAL: NCT02887521
Title: Pulmonary Rehabilitation Before Lung Cancer Resection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: A221502; NCI-2016-01105 (Registry Identifier: NCI Clinical Trial Reporting Program); NCT01682850 (obsolete NCT alias)
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pulmonary Disease, Chronic Obstructive | interventions — Educational Status; Rehabilitation; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Rehabilitation (PR) (Experimental): Patients will receive 10 in-clinic sessions of preoperative Pulmonary Rehabilitation (PR) two weeks prior to surgery. Patients will receive a Participant Manual demonstrating and explaining the rehabilitation process. Patients will also receive a log for recording their efforts and notes for every day until the day of surgery. A video recording of the intervention from start to finish will be provided to all patients. The video recording should be played in all 10 sessions at the registering site. The PR sessions will include breathing awareness, upper and lower extremity exercise, instructions for inspiratory muscle training using the PFlex valve, practice at home and goal setting. Patients undergo surgery and will be followed until 6 months following surgery. Patients complete follow up questionnaires at 3 and 6 months after discharge.
  Interventions: Other: education; Procedure: rehabilitation; Procedure: surgery
- Standard of Care (Active Comparator): Patients will receive a pedometer to monitor their daily steps and a pamphlet with exercises plus the standard course of care for patients undergoing lung resection surgery. The patients will not be asked to return the pedometer. The local institutional coordinator will go over the use of the pedometer and the exercise materials with the patient. The patients will be asked to keep a log of their pre-operative steps and mail the log to the registering site. Patients undergo surgery and will be followed until 6 months following surgery. Patients complete follow up questionnaires at 3 and 6 months after discharge.
  Interventions: Device: pedometer; Other: education; Procedure: surgery

INTERVENTIONS:
Other: education — pulmonary rehabilitation participant manual
  Arms: Pulmonary Rehabilitation (PR)
Procedure: rehabilitation — pulmonary rehabilitation
  Arms: Pulmonary Rehabilitation (PR)
Device: pedometer — receive a pedometer
  Arms: Standard of Care
Other: education — receive a pamphlet with exercises plus the standard course of care
  Arms: Standard of Care
Procedure: surgery — patients undergo surgery

SUMMARY:
This is a study funded by the National Institute of Health. The rationale for the need of this research is the lack of any well proven risk-reducing intervention that may decrease the morbidity of lung cancer resection in patients with COPD or that may improve their quality of life trajectory, a meaningful outcome in the overall disease progression. The proposed intervention is unique as it combines exercise and behavioral interventions that were pilot tested in a randomized single-blinded controlled design in the proposed population and proved feasible and potentially effective. The aim is to test the effect of the proposed rehabilitation on length of stay, pulmonary complications and quality of life trajectory.

DETAILED DESCRIPTION:
Prospectively, 194 patients will be randomized to either ten sessions of preoperative pulmonary rehabilitation (PR) vs. standard care at a number of healthcare centers throughout the United States. This study will be open for 36 months. Randomization will be stratified by three variables: very severe lung function (yes vs. no), prior neo-adjuvant chemotherapy for this operation (yes vs. no) and open thoracotomy vs. video assisted thoracoscopy. The primary and secondary objectives are provided below.

Primary Objective:

To prospectively determine the effect of 10 sessions of customized preoperative PR on the length of hospital stay in patients that undergo a lung cancer resection and have COPD compared to a matched control group. Hypothesis: Ten sessions of customized preoperative PR will significantly reduce the length of hospital stay.

Secondary Objectives:

1. To prospectively determine the effect of 10 sessions of customized preoperative PR on the number of postoperative complications in patients that undergo a lung cancer resection and have COPD compared to a matched control group.

   * Hypothesis: Ten sessions of customized preoperative PR will significantly reduce the number of postoperative pulmonary complications.
2. To prospectively determine the effect of a 10-session preoperative PR on the trajectory of quality of life at 3 and 6 months after the curative resection compared to a matched control group.

   * Hypothesis: Ten sessions of customized preoperative PR will significantly and meaningfully (more than the minimal clinically important difference) improve quality of life after surgery compared to a control group.

Patients will be followed at 3 and 6 months post-surgery.

ELIGIBILITY:
1. Patient is scheduled to undergo NSCLC resection: video assisted thoracoscopy (VATS) or open thoracotomy for: limited resection, lobectomy, or pneumonectomy. Surgery must not be scheduled to take place < 3 weeks after registration.
2. Patient has a doctor diagnosis of COPD.
3. Patient is a current or ex-smoker with a smoking history of ≥ 10 pack years. (Calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked. For example, 1 pack-year is equal to smoking 20 cigarettes (1 pack) per day for 1 year, or 40 cigarettes per day for half a year, and so on).
4. Age ≥ 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Benzo, MD, MSc, Study Chair — Mayo Clinic
Locations (7):
- United States (6):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Baylor University Medical Center, Dallas, Texas
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
- London Regional Cancer Program, London, Ontario, Canada

REFERENCES:
- [Derived] Perrotta F, Cennamo A, Cerqua FS, Stefanelli F, Bianco A, Musella S, Rispoli M, Salvi R, Meoli I. Effects of a high-intensity pulmonary rehabilitation program on the minute ventilation/carbon dioxide output slope during exercise in a cohort of patients with COPD undergoing lung resection for non-small cell lung cancer. J Bras Pneumol. 2019 Oct 14;45(6):e20180132. doi: 10.1590/1806-3713/e20180132. eCollection 2019. PMID 31618297

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pulmonary Rehabilitation (PR) | Standard of Care
Started | 4 | 5
Completed | 4 | 2
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Population: All patients that began protocol intervention were included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulmonary Rehabilitation (PR) | Standard of Care | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Median (Full Range); unit: years] | 69.5 [56 to 82] | 77 [73 to 86] | 75 [56 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 1 | 1
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay Assessed With Complete Admission Hospital Records
Description: The coordinator at each site will be responsible for sending complete de-identified hospital records from each patient to Dr. Benzo's staff, where a nurse blinded to the study arm will abstract the main outcome (length of stay and postoperative complications).
  The primary endpoint will be assessed at Dr. Benzo's office (Mayo Clinic) with the complete admission hospital records in order to extract the length of stay. The records will be mailed from the sites to Johanna Hoult in a pre-stamped envelope.
Time Frame: Up to 6 months
Population: Original plan for abstracting length of hospital stay from medical records did not occur due to study termination
Arm/Group | Pulmonary Rehabilitation (PR) | Standard of Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Post-operative Pulmonary Complications Assessed by Chart Review
Description: The following events will be considered postoperative pulmonary complications: pneumonia (new infiltrate + either fever (>38.5 C) and white cell count >11,000 or fever and purulent secretions), severe atelectasis (requiring bronchoscopy), prolonged chest tubes (>6 days), and respiratory failure (intubation or prolonged mechanical ventilation (>24 hours). These outcomes will be obtained by chart review by a nurse trained in the abstraction of the desired outcomes from the medical records and blinded to treatment assignment.
Time Frame: Up to 6 months
Population: Original plan for abstracting post-operative complications manually from medical records did not occur due to study termination.
Arm/Group | Pulmonary Rehabilitation (PR) | Standard of Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quality of Life (QOL) Assessed by Chronic Respiratory Questionnaire
Description: Chronic Respiratory Questionnaire (CRQ) (four domains: dyspnea, fatigue, emotional function and mastery). This instrument will be the primary tool to assess QoL given that it was specifically designed for COPD. Specifically, the CRQ represents one of the most well known, widely-applied, and psychometrically-sound patient reported outcomes for use in clinical trials involving patients with COPD. Each domain includes 4 to 7 items, with each item graded on 7-point Likert scale; item scores within a domain are summated to provide a total score for each domain. The endpoint value is the 6 month values minus the baseline values. Therefore the endpoint score may range from minus-7 to 7. Higher scores indicate better HRQL. A negative change from baseline to study completion indicates a worsening score.
Time Frame: At baseline and at 6 months
Population: All patients who registered and completed the CRQ at baseline and study completion were included in this analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pulmonary Rehabilitation (PR) | Standard of Care
Number analyzed (Participants) | 4 | 3
units on a scale
  Change in CRQ Dyspnea | 0.0 [-0.9 to 0.4] | -.6 [-1.4 to 0.5]
  Change in CRQ Fatigue | 1.0 [-2.0 to 4.3] | 1.5 [1.0 to 1.5]
  Change in CRQ Emotional function | 0.8 [-0.7 to 4.3] | 0.7 [0.3 to 2.0]
  Change in CRQ Mastery | 0.7 [-1.0 to 2.7] | 0.3 [-0.3 to 0.8]

4. Secondary Outcome: Quality of Life (QOL) Assessed by Linear Analog Self-Assessment
Description: LASA (single-item numerical analogue quality of life Questionnaire) individual QOL domain scores have been validated previously for lung cancer patient populations and for assessment of patient-reported outcomes in similar trials. Survey is based on 6 questions that are scored on a 0-10 scale with 0 being "as bad as it can be" and 10 being "As good as it can be." A negative change in score from baseline indicates a worsening score.
Time Frame: Up to 6 months
Population: Original plan for collecting and analyzing this data did not occur due to study termination
Arm/Group | Pulmonary Rehabilitation (PR) | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: We do not anticipate any adverse events related to participation in this study. PR has no reported risks based on 3000 patients with severe COPD in the National Emphysema treatment trial that underwent exercise training in more intensity compared to the one planned in this study. Therefore, no adverse events assessment were collected per protocol.
Description: We do not anticipate any adverse events related to participation in this study. PR has no reported risks based on 3000 patients with severe COPD in the National Emphysema treatment trial that underwent exercise training in more intensity compared to the one planned in this study. Therefore, no adverse events assessment were collected per protocol.
Arm/Group | Pulmonary Rehabilitation (PR) | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT02887521/Prot_SAP_ICF_000.pdf